CLINICAL TRIAL: NCT00385541
Title: The Comparison of Morphine and Hydromorphone Patient-Controlled Analgesia
Brief Title: Comparison of Side Effects of Morphine and Hydromorphone Patient-Controlled Analgesia (PCA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Pamela Flood, Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAA2949
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Results first posted 2010-08-31 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Post Operative Pain
Keywords: pain; morphine; hydromorphone; nausea; vomiting; pruritis
MeSH Terms: conditions — Pain, Postoperative; Pain; Nausea; Vomiting; Pruritus | interventions — Morphine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator): Patients receive morphine 1mg/dose PCA for postsurgical pain; max 10 mg/hr; lockout 6 minutes.
  Interventions: Drug: Morphine PCA
- B (Active Comparator): Patients receive hydromorphone 0.2mg/dose PCA for postsurgical pain; max 10mg/hr; lockout 6 minutes.
  Interventions: Drug: Hydromorphone PCA

INTERVENTIONS:
Drug: Morphine PCA — Morphine 1mg/mL, dose 1mL, lockout 6 minutes, max 10mL
  Other Names: Astramorph PF; Duramorph; Infumorph
  Arms: A
Drug: Hydromorphone PCA — hydromorphone PCA 0.2mg/lml, dose 1ml, lockout 6min, max 10ml
  Other Names: Dilaudid
  Arms: B

SUMMARY:
Both morphine and hydromorphone are pain medications commonly used after surgery. It is thought at the institution that hydromorphone causes less side effects but this has not been studied. The study proposes to treat the patients with either morphine or hydromorphone and determine how much nausea, vomiting, and itching they have with each drug

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for abdominal surgery requiring post-operative PCA
* ASA = I or II

Exclusion Criteria:

* preoperative pain or use of pain medication
* narcotic allergy
* morbid obesity (Body Mass Index > 30)
* diagnosis of sleep apnea
* hepatic or renal disease
* use of medications that would affect narcotic pharmacodynamics
* preoperative nausea, vomiting, or pruritis
* diagnosis of alcoholism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2003-11 (Actual); Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Flood, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Result] Hong D, Flood P, Diaz G. The side effects of morphine and hydromorphone patient-controlled analgesia. Anesth Analg. 2008 Oct;107(4):1384-9. doi: 10.1213/ane.0b013e3181823efb. PMID 18806056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults having general surgery at Columbia University Medical Center (CUMC) were randomly assigned to receive Patient-Controlled Analgesia (PCA) with morphine or hydromorphone
Pre-assignment Details: Double blind randomized controlled trial. Patients under 18, with chronic pain or on pain medication before surgery were excluded.
Groups:
- Morphine PCA: Patients receive morphine 1mg/dose pca for postsurgical pain. Max 10mg/hr, lockout 6 minutes
- Hydromorphone PCA: Patients receive hydromorphone via PCA at 0.2mg/dose, max 2mg/hr lockout 6 minutes
Period: Overall Study
Arm/Group | Morphine PCA | Hydromorphone PCA
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — severe pain, clinician requested unblind | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine PCA | Hydromorphone PCA | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12) | 44 (8) | 42.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Nausea Assessment by Patient
Description: Nausea scale range: (0 = none, 10 = the worst), ordinal.
Time Frame: 1 hour after surgery, 8 hours after surgery
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Morphine PCA | Hydromorphone PCA
Number analyzed (Participants) | 25 | 25
Units on a scale | 4.6 (3.2) | 3.0 (2.5)

2. Secondary Outcome: Mean Score on the Numeric Rating Scare (NRS) Pruritus Scale
Description: The NRS Pruritus Scale was used to measure magnitude of pruritus (0 = none, 10 = the worst).
Time Frame: 1 hour after surgery, 8 hours after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Morphine PCA | Hydromorphone PCA
Number analyzed (Participants) | 25 | 25
Units on a scale | 2 (0) | 2.5 (1.3)

3. Secondary Outcome: Pain Assessment by Patient
Description: Numeric Rating Scale for Pain: (0 = none, 10 = the worst), ordinal.
Time Frame: 1 hour after surgery, 8 hours after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Morphine PCA | Hydromorphone PCA
Number analyzed (Participants) | 25 | 25
Units on a scale | 7.9 (2.3) | 7.1 (2.4)

4. Secondary Outcome: The Number of Patients Who Vomited
Time Frame: 1 hour after surgery, 8 hours after surgery
Measure: Number; unit: participants
Arm/Group | Morphine PCA | Hydromorphone PCA
Number analyzed (Participants) | 25 | 25
participants | 1 | 0

5. Secondary Outcome: Mean Score on the Ramsey Scale of Sedation
Description: The Ramsey scale is used as a measure of sedation from 1 (the patient in anxious and agitated) to 6 (the patient exhibits no response).
Time Frame: 1 hour after surgery, 8 hours after surgery
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Morphine PCA | Hydromorphone PCA
Number analyzed (Participants) | 25 | 25
score on scale | 2.8 (0.6) | 2.8 (0.7)

ADVERSE EVENTS:
Arm/Group | Morphine PCA | Hydromorphone PCA
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
This was a small study under typical clinical conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No